CLINICAL TRIAL: NCT00032916
Title: Drug Interaction Study With NS2359 and Cocaine in Cocaine Experienced Volunteers
Brief Title: Drug Interaction Study With NS2359 and Cocaine in Cocaine Experienced Volunteers - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-2359-02-1; NCT00031330 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2004-04

CONDITIONS: Cocaine-Related Disorders; Drug Administration Schedule; Infusions, Intravenous
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — GSK372475

INTERVENTIONS:
Drug: NS2359

SUMMARY:
The purpose of this study is to conduct a drug interaction study with NS2359 and cocaine in cocaine experienced volunteers.

DETAILED DESCRIPTION:
This is a single-center, double-blind, placebo-controlled, randomized, single dose, fixed order, dose escalating inpatient design that will study oral NS2359 in cocaine experienced volunteers.

ELIGIBILITY:
Inclusion Criteria:

Male or Female, 18-45 yrs of age; females of child-bearing potential using appropriate method of birth control; be able to understand the procedure and agrees to participate via informed consent; must be cocaine dependent according to DSM-4 criteria; must be capable of providing written consent; must be able to comply with protocol requirement, CPU rules and regulations; must not be currently seeking treatment for cocaine abuse.

Exclusion Criteria:

Incapable of understanding the informed consent process; Additional criteria available during screening at the site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2001-06; Study Completion 2002-12

PRIMARY OUTCOMES:
Pharmacokinetic parameter comparison
plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States